CLINICAL TRIAL: NCT07123961
Title: Pediatric Acute Respiratory Distress Syndrome (ARDS) Management (PARMA) Trial
Brief Title: Pediatric Acute Respiratory Distress Syndrome (ARDS) Management Trial
Acronym: PARMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-022470
Record Dates: First submitted 2025-08-06; First posted 2025-08-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Ventilator Management; Lung-protective Ventilation; Pediatric Acute Respiratory Distress Syndrome (PARDS)
Keywords: Acute Respiratory Distress Syndrome; ARDS; Vent; Ventilator; Ventilator Management; Pediatric ARDS; Pediatric Ventilator Management; PARDS; Pediatric ARDS Protocolized Treatment; Invasive Mechanical Ventilation; IMV; Pediatric Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible and consented subjects will be randomized within 24 hours of meeting study eligibility using 1:1 permuted blocks, using a randomization module available in Research Electronic Data CAPture (REDCap).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Driving Pressure Mechanical Ventilation (Active Comparator): A participant who is already on the breathing machine will have the driving pressure set to 25 cmH2O (rate of pressure delivery). All other standard clinical care for this participant will stay the same based on what their clinical team chooses to do.
  Interventions: Other: High Driving Pressure Mechanical Ventilation
- Low Driving Pressure Mechanical Ventilation (Active Comparator): A participant who is already on the breathing machine will have the driving pressure set to 15 cmH2O (rate of pressure delivery). All other standard clinical care for this participant will stay the same based on what their clinical team chooses to do.
  Interventions: Other: Low Driving Pressure Mechanical Ventilation

INTERVENTIONS:
Other: High Driving Pressure Mechanical Ventilation — A participant who is already invasively mechanically ventilated will be placed on "Pressure Control Ventilation" mode on an Evita V500 (Manufacturer: Dräger, Lübeck, Germany) ventilator if they are not already. The driving pressure will be set to 25 cmH2O (rate of pressure delivery). The Children's Hospital of Philadelphia (CHOP) PICU's standard of care regarding sedation, fluid management, ventilator weaning, and extubation readiness for invasively mechanically ventilated children will be adhered to for the duration of the study. An Enlight 2100 Electrical Impedance Tomography (EIT) Device (Manufacturer: Timpel) strap will be placed across the participant's chest up to four times throughout the study for a few hours to image the aeration in the lungs.
  Arms: High Driving Pressure Mechanical Ventilation
Other: Low Driving Pressure Mechanical Ventilation — A participant who is already invasively mechanically ventilated will be placed on "Pressure Control Ventilation" mode on an Evita V500 (Manufacturer: Lübeck, Germany) ventilator if they are not already. The driving pressure will be set to 15 cmH2O (rate of pressure delivery). CHOP PICU's standard of care regarding sedation, fluid management, ventilator weaning, and extubation readiness for invasively mechanically ventilated children will be adhered to for the duration of the study. An Enlight 2100 (EIT) Device (Manufacturer: Timpel) strap will be placed across the participant's chest up to four times throughout the study for a few hours to image the aeration in the lungs.
  Arms: Low Driving Pressure Mechanical Ventilation

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a serious and potentially life-threatening lung condition that can affect children. Currently, ventilator settings commonly used in treatment are based on approaches developed for adults, and it remains unclear whether these settings are equally effective for children. Because children's bodies respond differently than adults', it is important to determine the most effective ventilator strategies specifically for pediatric patients. This study will compare two different ventilator approaches in children with ARDS to identify which method provides the greatest benefit. The findings will also help inform the design of a larger study in the future.

ELIGIBILITY:
Inclusion:

1. age > 2 weeks (> 38 weeks corrected gestational age) and < 18 years (not yet had 18th birthday)
2. acute (≤ 7 days of risk factor) respiratory failure requiring invasive mechanical ventilation
3. ventilated with endotracheal tube or tracheostomy for ≤ 7 days from risk factor onset
4. hypoxemia defined as PaO2/FIO2 (measurement of the amount of oxygen dissolved in the blood plasma/concentration of inhaled oxygen) > 300 (or SpO2/FIO2 (measurement of the percentage of hemoglobin in your blood that is carrying oxygen/concentration of inhaled oxygen) > 315 on Positive End-Expiratory Pressure (PEEP) ≥ 5 cmH2O (rate of pressure delivery) on two consecutive measurements 4 hours apart and sustained at the time of consent and randomization
5. bilateral opacities on chest radiograph as determined by radiologist, clinical attending, or PI

Exclusion:

1. hypoxemia caused primarily by hydrostatic pulmonary edema from heart failure or fluid overload
2. non-palliated or unrepaired cyanotic congenital heart disease
3. ventilated via tracheostomy at baseline prior to acute illness
4. obstructive airway disease determined to be the primary cause of respiratory failure
5. severe moribund state not expected to survive > 72 hours
6. any limitations of care at time of screening
7. escalation to high frequency oscillatory ventilation or extracorporeal support (i.e., meeting PARMA protocol failure criteria) at time of screening
8. previous enrollment in this study

Ages: 38 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Sustained Resolution of Hypoxemia | Up to 672 hours
  The primary outcome of PARMA is time (in hours) per participant to sustained resolution of hypoxemia, defined as being alive with PaO2/FIO2 (measurement of the amount of oxygen dissolved in the blood plasma/concentration of inhaled oxygen) > 300 (or SpO2/FIO2 (measurement of the percentage of hemoglobin in your blood that is carrying oxygen/concentration of inhaled oxygen) > 315) on two consecutive measurements 4 hours apart. This outcome is censored at 28 days (672 hours).

SECONDARY OUTCOMES:
Imaging (Electrical Impedance Tomography (EIT)): Lung recruitment | Once from time of enrollment to randomization, once within 8 hours post-randomization and once within 24-72 hours after randomization.
  EIT (Electronic Impedance Tomography) is an FDA-approved non-radiating method of imaging lung aeration. EIT bands are placed on the subject and EIT imaging will be performed at three time points to assess the assigned study arm. The percentage of patients with recruited lung at the immediate post-randomization EIT, relative to pre-randomization EIT measurement will be determined.
Imaging (Electrical Impedance Tomography (EIT)): Overdistension | Once from time of enrollment to randomization, once within 8 hours post-randomization and once within 24-72 hours after randomization.
  EIT (Electronic Impedance Tomography) is an FDA-approved non-radiating method of imaging lung aeration. EIT bands are placed on the subject and EIT imaging will be performed at three time points to assess the assigned study arm. The percentage of patients with overdistended lung at the immediate post-randomization EIT, relative to pre-randomization EIT measurement will be determined.
Imaging (Electrical Impedance Tomography (EIT)): Center of Ventilation | Once from time of enrollment to randomization, once within 8 hours post-randomization and once within 24-72 hours after randomization.
  EIT (Electronic Impedance Tomography) is an FDA-approved non-radiating method of imaging lung aeration. EIT bands are placed on the subject and EIT imaging will be performed at three time points to assess the assigned study arm. The average value of center of ventilation for each study arm at the immediate post-randomization EIT will be compared.
Clinical End Point: all-cause mortality at 90 days | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants all-cause mortality at 90 days after enrollment or hospital discharge.
Clinical End Point: all-cause mortality at 28 days | From enrollment up to hospital discharge, no longer than 28 days.
  Total number of participants all-cause mortality at 28 days after enrollment or hospital discharge.
Clinical End Point: Pediatric ICU discharge | From enrollment up to pediatric ICU discharge, no longer than 90 days
  Total days per participant until Pediatric ICU discharge from start of enrollment.
Clinical End Point: Hospital Discharge | From enrollment up to hospital discharge, no longer than 90 days.
  Total days per participant until hospital discharge from enrollment.
Clinical End Point: Primary Cause of Death | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants who meet primary cause of death as defined as brain death, other neurologic, multiple organ dysfunction syndrome, refractory shock, refractory hemorrhage or refractory hypoxemia.
Clinical End Point: Ventilator Free Days | From enrollment up to hospital discharge, no longer than 28 days.
  Total ventilator free days (VFDs) per participant at 28 days (defined as number of days alive and off invasive ventilation by day 28).
Clinical End Point: New Oxygenation- or Ventilator-dependency | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants with new oxygenation- or ventilator-dependency at time of discharge.
Safety Endpoint: pneumothorax requiring chest tube | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants with diagnosis of pneumothorax requiring chest tube.
Safety Endpoint: other air leak not requiring chest tube | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants with diagnosis of other air leak not requiring chest tubes.
Safety Endpoint: ventilator-associated pneumonia | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants with diagnosis of ventilator-associated pneumonia.
Safety Endpoint: new or progressive multiple organ dysfunction syndrome | From enrollment up to hospital discharge, no longer than 90 days.
  Total number of participants with diagnosis of new or progressive multiple organ dysfunction syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Nadir Yehya, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified trial dataset, stripped of all personal health information, will be shared with an existing NIH data repository (likely the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH)).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data (IPD) will be shared 1 year after main manuscript publication.
Access Criteria: The IPD will be made readily available for research by qualified individuals within the scientific community as determined by DASH's regulatory and contractual requirements. The dataset will be accessible via the DASH platform.

DOCUMENTS (2):
  • Study Protocol (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT07123961/Prot_000.pdf
  • Informed Consent Form (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT07123961/ICF_001.pdf